CLINICAL TRIAL: NCT00452998
Title: Sequential Laser Iridotomy Using Argon and Q-Switched 532 nm Frequency Doubled Neodymium Yag Laser: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Cecilia Aquino, MD, National University Hospital, Singapore
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSRB A/06/293
Record Dates: First submitted 2007-03-27; First posted 2007-03-28 (Estimated); Last update posted 2008-05-14 (Estimated); Status verified 2008-05

CONDITIONS: Chronic Angle Closure Glaucoma; Primary Angle Closure; Primary Angle Closure Suspect; Fellow Eyes of Acute Angle Closure Glaucoma
Keywords: Sequential Laser Iridotomy; Q-Switched 532 nm Laser; Frequency Doubled Neodymium Yag Laser

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Q-switched fd Nd:yag in Laser Iridotomy

SUMMARY:
Sequential Laser Iridotomy uses argon and Nd:yag laser in the first and second steps, respectively. Using q-switched 532 nm laser in the second step is hypothesized to be as good and effective as the conventional Nd:yag laser, because it selectively targets pigmented cells and delivers a short pulse duration of 3 nanoseconds, causing less thermal and collateral damage.

DETAILED DESCRIPTION:
Laser iridotomy is an established procedure in the management of angle closure glaucoma (ACG) and for prophylaxis in the fellow eyes.

Sequential argon-YAG (SAY) laser iridotomy is the serial use of argon and Nd:YAG laser at the same treatment session to create an iridotomy. Argon laser is initially used to make a bore of about 500 μm in diameter to an estimated two-thirds iris thickness in depth. The 1064 nm Q-switched neodymium YAG laser is next used to complete the perforation1. Others aim the argon laser at the iris surface to create a crater, and the next shots at the base of the crater until the iris is penetrated as evidenced by a pigment plume. The Nd:YAG laser then creates a photodisruptive explosion to enlarge the opening.

This procedure was first described by Zborwski-Gutman in 1988. Sixteen eyes were treated with two argon stretch burns and up to 35 penetrating burns that produced an iridotomy that was either imperforate or inadequate. Nd:YAG laser was used to complete the iridotomy. In all the eyes, the iridotomy was achieved in one session, and two eyes had a moderate increase in pressure that was easily controlled. The authors found that the total energy levels for each laser modality were significantly lower than those previously reported using either laser alone. The authors concluded that the sequential technique is safe and effective, and is recommended for iridotomy in difficult iris types.

Lim et al in 1996 did a prospective study that compared argon laser iridotomy and SAY in dark irides. Twenty-four eyes of 17 patients were involved; and 13 underwent argon laser iridotomies, and 11 underwent SAY. The argon laser settings were standardized at 1.2 W, 50 μm spot size and 0.1 second duration. The Nd: YAG laser was set at 2.5 mJ and single-pulse shots were used. All the iridotomies were completed in a single session. The mean total energy used for argon laser iridotomy was 8.28 J; while for SAY, 3.12 J was used for the argon laser stage and 7.5 mJ for the Nd:YAG stage. The authors concluded that the total argon laser energy used can be reduced by 2.65 times using the SAY technique.

The SAY technique is ideal in Asian eyes because it avoids the disadvantages of argon and Nd-YAG laser, when they are used as separate methods.

In SAY, bleeding is uncommon and microscopic, unlike in Nd:YAG iridotomy wherein it can be severe enough to cause the abortion of the procedure. Nd:YAG iridotomy is rarely associated with focal lens or retina damage; but argon laser can cause inadvertent focal lens damage.

By using ND:YAG laser as second stage laser, SAY iridotomy avoids the tedious and hazardous chipping enlargement phase of argon iridotomy that can contribute to retinal damage. Likewise, with the argon laser pre-treatment, excessive pigment and debris dispersion, iris splintering, and high energy levels needed for iris perforation from a Nd:YAG iridotomy in an Asian eye is avoided. In Ho's series of 20 patients who underwent SAY, only one eye had iridotomy closure during a mean follow-up period of 14 months.

Q-switched 532 nm frequency-doubled neodymium:yytrium-aluminum-garnet (fd-Nd:YAG) laser has been used in the recent years for selective laser trabeculoplasty (SLT). It was developed by Latina et.al. to selectively target pigmented trabecular meshwork (TM) cells without causing thermal or collateral damage to the nonpigmented cells or structures of the TM. This is so because it is able to deliver a short pulse duration of 3 nanoseconds while selectively lysing intracellular melanosomes, killing pigmented cells and leaving cellular membranes and neighboring nonpigmented cells intact. This technique delivers less than 1% of the energy of ALT, with shorter pulse durations and consequently higher power levels. Latina noted bubble formation at higher fluence, but this is not from boiling tissue, but are microcellular cavitation effects.

ELIGIBILITY:
Inclusion Criteria:

* More than 21 years old
* Able to give informed consent
* Diagnosis of either: chronic angle closure glaucoma (CACG), primary angle closure (PAC), primary angle closure suspect (PACS) or fellow eyes of acute angle closure glaucoma (AACG), and in need of a laser iridotomy

Exclusion Criteria:

* History of any prior laser treatment or intraocular surgery to the eye
* History of any corneal disease
* Any ocular infection/ inflammation within the last two months
* Inability to give informed consent

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2006-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Visual Acuity
Intraocular pressure
Total power delivered by each laser modality
Iridotomy patency and size
Pain rating during the procedure
Anterior segment inflammation
Endothelial cell count
Cataract progression
Rate of complications

CONTACTS AND LOCATIONS:
Overall Officials: Paul Chew, FRCSEd,MMed, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Latina MA, Park C. Selective targeting of trabecular meshwork cells: in vitro studies of pulsed and CW laser interactions. Exp Eye Res. 1995 Apr;60(4):359-71. doi: 10.1016/s0014-4835(05)80093-4. PMID 7789416